CLINICAL TRIAL: NCT06160284
Title: Exploration of Synaptotrophic Effects of Psilocybin in Opioid Use Disorder (OUD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000036178; P30DA046345 (NIH)
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Participants will be medically healthy females and males with OUD.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Current OUD diagnosis + psilocybin (Experimental): All participants will receive a [11C]-UCB-J PET scan and fMRI with in 1-2 weeks pre and post treatment with one dose of Psilocybin. Intravenous lines will be used for phlebotomy and administration of the [11C]-UCB-J radiotracer. On the PET scanning day, a radial arterial catheter may be inserted.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a single dose of psilocybin administered in 20 mg or 25 mg doses depending on the participant's weight: 20 mg (among participants < 70 kg) or 25 mg (among participants >70 kg). Participants will be administered psilocybin at CNRU, within 1-2 weeks of the baseline [11C]-UCB-J PET.

SUMMARY:
This study will examine the synaptotrophic effects of psilocybin among medically healthy, detoxified OUD subjects. Eligible OUD participants will undergo pre- and post- psilocybin administration PET scans with the [11C]-UCB-J radiotracer while inpatient.

DETAILED DESCRIPTION:
Participants will undergo screening as outpatients at the Clinical Neuroscience Research Unit (CNRU). Once deemed eligible, OUD subjects will be studied as inpatients. However, they will have the option of scheduling their second [11C]-UCB-J PET as an outpatient (pending these participants' agreement to undergo outpatient visits twice per week to provide urine toxicology to monitor abstinence before PET).

The only portion of the study that will be available as outpatient for OUD subjects will be the 1-2 weeks before the second [11C]-UCB-J PET scan. The subject will still be admitted for 1-2 weeks, which will include: inpatient detoxification, baseline [11C]-UCB-J PET scan, psilocybin administration, and overnight observation after psilocybin administration. However, they may be discharged the day following psilocybin administration and return 2x weekly for urine toxicology testing between discharge and the second [11C]-UCB-J PET to confirm abstinence.

Structural magnetic resonance imaging (MRI) scans will be obtained for anatomical registration/partial volume correction from all subjects. Functional MRI (fMRI) scans will be completed pre- and post-psilocybin administration to evaluate changes in resting state connectivity. All subjects will participate in a battery of behavioral assessments for exploratory correlations with [11C]-UCB-J. Inpatient subjects who smoke cigarettes will have the option of using nicotine gum and/or nicotine patch while on the unit in order to prevent or minimize nicotine withdrawal. The [11C]-UCB-J PET scans will be done at the Yale PET Center 1-2 weeks before (baseline) and after psilocybin administration.

This is a single-center study at Yale, that will have study activities completed at the following areas:

* Clinical Neuroscience Research Unit (CNRU) of the Connecticut Mental Health Center (CMHC)
* Yale Positron Emission Tomography (PET) Imaging Center
* Yale Magnetic Resonance Research Center (MRRC)

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written, informed consent;
* Physically healthy by medical history, physical, neurological, ECG, and laboratory examinations;
* DSM-5 criteria for Opioid Use Disorder;
* Documented evidence (by urine toxicology) of opioid use (upon screening);
* Inpatient verified > 1 week of abstinence;
* For females, a negative serum pregnancy (beta-HCG) test.

Exclusion Criteria:

* DSM-5 criteria for other substance use disorders (e.g., alcohol, cocaine, sedative hypnotics), except for nicotine (concurrent alcohol or drug use is allowed if it does not meet criteria for a substance use disorder and does not take place during inpatient stay)
* A primary DSM-5 Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression, as determined by psychiatric history (Mini International Neuropsychiatric Interview, MINI), or another disorder that may interfere with the study's primary outcomes in the view of PI
* Immediate (first-degree relative) family history of formally diagnosed schizophrenia or other psychotic disorders (e.g., delusional disorder, schizoaffective disorder), or bipolar I/II disorder
* A history of significant and/or uncontrolled medical or neurological illness
* Hypertension at screening defined as: systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg;
* History of cardiovascular disease, including but not limited to clinically significant coronary artery disease, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, angina pectoris, coronary artery bypass graft or artificial heart valve, stroke, transient ischemic attack, or any clinically significant arrhythmia
* Any clinically significant abnormal electrocardiogram (ECG) finding, such as findings suggestive of ischemia or infarct, complete bundle branch block, atrial fibrillation or other symptomatic arrhythmia, or predominantly non-sinus rhythm, at screening
* Resting QT interval with Fridericia's correction (QTcF) ≥ 450 msec (male) or ≥ 470 msec (female) at Screening, or inability to determine QTcF interval
* Presence of risk factors for torsades de pointes, including: long QT syndrome, uncontrolled hypokalemia or hypomagnesemia, history of cardiac failure, history of clinically significant/symptomatic bradycardia, family history of idiopathic sudden death or congenital long QT syndrome, or concomitant use of a torsadogenic medication
* Current use of psychotropic and/or potentially psychoactive prescription medications considered to the investigators are likely to interfere clinically with human subject's safety (i.e., contraindicated drug-drug interactions with psilocybin) or scientifically (i.e., likely to influence or alter outcomes of the study)
* Medical contraindications to MRI procedures (e.g., ferromagnetic implants/foreign bodies, claustrophobia, etc.)
* Arterial Line Exclusion: Blood donation within eight weeks of the start of the study
* Arterial Line Exclusion: History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto)
* Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits followed by the Yale PET Center (21CFR361.1).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Synaptic Density | baseline and 1-2 weeks post treatment
  Change in synaptic density pre- and post- psilocybin administration will be measured using [11C]-UCB-J PET (volume of distribution [VT] and binding potential [BPND]) among OUD. The regions of interest (ROI) will be subregions of the prefrontal cortex identified by preclinical and preliminary clinical studies.
Association between VT and BPND | up to 12 weeks
  Association between VT and BPND assessed to determine whether changes in VT are associated with changes in BPND.
Time to relapse | up to 12 weeks
  Mean number of days to relapse assessed by self- report
Urine toxicology post treatment | up to 12 weeks
  The mean number of positive urine tests post treatment will be assessed. Urine samples will be tested for the presence of opioids. A positive test indicates opioid usage in the last 2 weeks.

SECONDARY OUTCOMES:
Change in vital signs- heart rate (HR) | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in heart rate measured in beats per minute during Psilocybin session
Change in vital signs- respiratory rate (RR) | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in respiratory rate measured in breaths per minute during Psilocybin session
Change in vital signs- oxygen saturation | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in percent oxygen saturation assessed using a pulse oximeter during Psilocybin session
Change in vital signs- systolic blood pressure | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in systolic blood pressure in mmHg during Psilocybin session
Change in vital signs- diastolic blood pressure | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in diastolic blood pressure in mmHg during Psilocybin session
Change in vital signs- body temperature | immediately prior to psilocybin treatment with and up to 5 hours+ post treatment
  Mean change in body temperature in degrees Fahrenheit during Psilocybin session
Total number of participants with treatment emergent adverse events | up to 12 weeks
  Total number of participants with any treatment emergent adverse events while on study assessed using the Systematic Assessment for Treatment Emergent Events (SAFTEE).
Change in Profile of Mood States (POMS) Score | approximately 30 and 150 minutes post Psilocybin treatment
  POMS is a validated 30 item questionnaire used to assess an individual's mood states. Total scores range from 0 to 120 with lower scores indicating a better mood state.
Change in Clinical Opioid Withdrawal Scale (COWS) Score | approximately 30 and 150 minutes post Psilocybin treatment
  COWS is an 11-item scale to rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score determines the stage/severity of opiate withdrawal and assess the level of physical dependence on opioids. Score: 5- 12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal
Change in Subjective Opioid Withdrawal Scale (SOWS) Score | approximately 30 and 150 minutes post Psilocybin treatment
  SOWS is a self-administered scale for opioid withdrawal symptoms. It has16 symptoms whose intensity is rated on a scale of 0 (not at all) to 4 (extremely). Mild Withdrawal = score of 1-10, Moderate withdrawal = 11-20, Severe withdrawal = 21-30
Change in Opioid Symptom Checklist (OSC) | approximately 30 and 150 minutes post Psilocybin treatment
  The OSC is a 13-item opioid symptom checklist consisting of true/false questions designed to measure opioid effects (e.g., "My skin is itchy"). True scores are totaled up to acute opiate positive and negative symptoms and low true scores will mean not feeling any of the negative and positive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Angarita, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes